CLINICAL TRIAL: NCT01517165
Title: Pioglitazone as an Aid During Buprenorphine Taper
Brief Title: Pioglitazone to Treat Opioid Withdrawal Symptoms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 999912469; 12-DA-N469
Record Dates: First submitted 2012-01-24; First posted 2012-01-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-02-02

CONDITIONS: Opioid-Related Disorders
Keywords: Opioid Dependence; Pioglitazone; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Pioglitazone

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: Pioglitazone
- Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone
  Arms: Group 1
Drug: Placebo
  Arms: Group 2

SUMMARY:
Background:

* Opioid-withdrawal symptoms include runny nose, body aches, chills, sweating, and diarrhea. Many people have these symptoms when trying to stop using opioid drugs. Long-acting opioids like methadone and buprenorphine are used to help people stop using other opioids, but these drugs can cause the same withdrawal symptoms. There are no non-opioid drugs that are approved specifically to treat those symptoms.
* Pioglitazone is a drug used to treat type 2 diabetes. In a research study, the drug allowed heroin users to decrease their methadone dose faster without much discomfort, and stay abstinent from heroin. Researchers want to learn more about how pioglitazone helps treat opioid withdrawal symptoms.

Objectives:

- To test whether pioglitazone can reduce opioid withdrawal symptoms.

Eligibility:

- Individuals between 18 and 65 years of age who will be using buprenorphine to treat opioid dependency.

Design:

* This study will last up to 17 weeks. Participants must come to the study clinic every day for at least 13 weeks.
* Participants will be screened with a physical exam and medical history. They will also answer questions about drug use habits, and provide blood and urine samples.
* Participants will take buprenorphine daily for 7 weeks. For the first 3 weeks, the dose will be increased to a level that should help stop the use of opioids. For the next 4 weeks, the dose will be decreased. Blood, urine, and breath samples will be collected at different study visits. Participants will also fill out questionnaires about mood, drug craving, and withdrawal symptoms.
* After 1 week on buprenorphine, participants will start the study pill (pioglitazone or a placebo) every day. They will take the study pill for 13 weeks.
* During the treatment period, participants will have drug counseling once a week for 30 minutes.
* Some participants have other tests as part of this study. These tests include functional magnetic resonance imaging scans to look for changes in brain activity and giving samples of cerebrospinal fluid to study brain chemistry.
* Participants will have a final followup phone call 3 weeks after the last clinic visit.

DETAILED DESCRIPTION:
Background:

Some individuals successfully maintained on buprenorphine or methadone are appropriate candidates for dose tapering and transition to medication-free follow-up care. For such individuals, the physical discomfort of the dose taper can be a barrier to a successful transition. Recent data suggest a novel approach: the FDA-approved diabetes medication pioglitazone (Actos), which activates the gamma (g) subtype of peroxisome-proliferator-activated receptors (PPARs). Pioglitazone acts not only in peripheral tissue, but also in brain regions associated with drug tolerance and withdrawal. In animal models, pioglitazone prevents signs of opioid withdrawal. In a small, preliminary open-label clinical study, opioid-maintained outpatients given pioglitazone were remarkably successful in transitioning comfortably to a medication-free state, after prior unsuccessful attempts without pioglitazone. These initial data provide proof of principle and indicate that pioglitazone merits evaluation in a randomized-controlled study.

Scientific goals:

(1) To determine whether, compared to placebo, pioglitazone increases successful completion of an opioid agonist/antagonist taper in patients who are physically dependent on opioids. (2) To determine the neural mechanisms by which such an effect may occur.

Participant population:

A total of up to 120 opioid-dependent participants (80 evaluable) will be enrolled. Evaluable participants are defined as those who are randomized to one of the two main experimental groups (pioglitazone or placebo). Target enrollment will include 25% women and 70% minorities (mostly African-American).

Experimental design and methods:

The study will be a randomized, double-blind clinical trial with two treatment groups (40 per group): pioglitazone (45 mg oral daily) and placebo. The study will last up to 10 weeks. All participants will receive 27 days of buprenorphine/naloxone (referred to hereinafter as buprenorphine) - 14 days of stabilization and a 13-day taper. Pioglitazone/placebo will be initiated in week 2 and continue for 5 weeks (3 weeks concurrently with buprenorphine and 2 weeks without). Participants will have two follow-up assessments: a clinic visit (week 7 or one week post-pioglitazone/placebo) and a phone follow-up (week 10 or 4 weeks post-pioglitazone/placebo). Participation will be conducted as a combination of outpatient and inpatient portions: first two weeks (pre-buprenorphine taper) as outpatients; 18 days on an inpatient unit (JHBC CRU) during and for approximately 5 days after the buprenorphine taper; and 10 daily visits and two follow-up visits outpatient. Throughout the study, participants will receive weekly individual counseling, including case management to prepare for post-study treatment. Data on opiate-withdrawal symptoms and craving will be collected daily. Data on self-reported drug use, with urine specimens for drug testing, will be collected three times weekly. A subset of participants will undergo functional magnetic-resonance imaging (fMRI) and magnetic-resonance spectroscopy (MRS): one training session in the mock scanner and two scanning sessions that will occur at the end of the first week of buprenorphine and during the second week of the buprenorphine taper. Another subset of participants (largely overlapping with the subset who undergo fMRI/MRS) will undergo one lumbar puncture so that we can measure levels of neurotransmitters, metabolites, and proinflammatory cytokines in cerebrospinal fluid (CSF). At the lumbar-puncture visit, blood will also be drawn so that we can compare analyte levels in CSF and blood. At the end of the study, all participants will be offered assistance to transfer to another treatment program, either drug-free treatment or opioid-agonist treatment (OAT). The primary outcome measures will be opioid-withdrawal severity as measured on the SOWs and COWs. Secondary outcome measures will include overall proportions of opioid-negative urines, proportions of participants needing adjunct medications, time to resumption of opioid use following discharge from the residential unit, status at follow-up, and (in the subset of participants who agree to undergo lumbar puncture) CSF levels (and corresponding blood levels) of proinflammatory cytokines and other analytes, which we hypothesize will predict outcome and thereby clarify pioglitazone s mechanism of action. In the subset of participants who agree to undergo fMRI/MRS and lumbar puncture, we will attempt to determine the neural mediators of pioglitazone s therapeutic effects, or (if pioglitazone is not effective) to determine predictors of treatment outcome. Post-treatment outcome measures are expected to be affected only indirectly by pioglitazone; we anticipate that pioglitazone will reduce withdrawal symptoms, enhance initial abstinence during the buprenorphine taper, and address possible protracted withdrawal.

Benefits to participants and/or society:

Participants will receive buprenorphine taper and drug counseling. There may be incidental benefits from the buprenorphine and counseling, because they are likely to reduce participants' use of opioids and risk of infectious diseases such as HIV or hepatitis B and C.

Risks to participants:

Participants may experience side effects from pioglitazone and/or buprenorphine/naloxone and are likely to experience some discomfort from opioid withdrawal. The subset of participants who agree to undergo lumbar puncture and fMRI/MRS may experience side effects from those procedures.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age between 18 and 65
  2. Evidence of physical dependence on opioids (determined by a combination of self-report, urine screen, and/or physical exam)
  3. Seeking detoxification treatment for opioid dependence
  4. Able to attend the clinic 7 days/week and undergo an 18-day residential stay
  5. For women:

     1. post-menopausal or surgically sterile (tubal ligation or hysterectomy) or
     2. if sexually active with a male partner and able to get pregnant, documented agreement to use an IRB-approved form of birth control. Acceptable forms of contraception for this study include: hormonal contraceptives (birth-control pills, injectable hormones, vaginal-ring hormones); IUD; diaphragm with spermicide; condom with spermicide.

EXCLUSION CRITERIA:

1. Any medical illness that in the view of the investigators would compromise participation in research (determined by Medical History; Physical Examination; Blood and Urine Laboratory tests; see details under Screening measures below), including, but not limited to:

   * Diabetes mellitus Type I or Type II
   * Past or current diagnosis of congestive heart failure
   * Signs and symptoms consistent with congestive heart failure including but not limited to fatigue, exercise intolerance, decreased peripheral perfusion, orthopnea, dyspnea on exertion, paroxysmal nocturnal dyspnea, peripheral edema, elevated jugular-venous pressure, pleural and pericardial effusions, hepatic congestion, ascites, elevated BUN and creatinine, hyponatremia, and elevated serum levels of hepatic enzymes.
   * Cardiovascular disease (e.g., history of congenital heart defect, heart disease, symptomatic coronary-artery disease, heart attack, irregular heartbeat, etc.)
   * Cerebrovascular disease
   * Unexplained history of syncope
   * History of seizures, except for febrile seizures at childhood
   * History of head injury with loss of consciousness of more than 30 minutes or with postconcussive sequelae lasting more than two days, regardless of loss of consciousness
   * Chronic renal failure as estimated by glomerular filtration rate (GFR) <60 mL/min/1.73 m(2)
   * CD4 < 200 or evidence of severely compromised immune system /AIDS
   * Active bladder cancer or history of bladder cancer
2. Allergy, hypersensitivity, or intolerance to buprenorphine, pioglitazone, other TZDs, or the metabolites of any of those drugs (determined by Medical History)
3. Pregnancy or breastfeeding (Urine Pregnancy Test; self-report)
4. Diabetes medications (e.g., sulfonylureas, metformin, insulin, etc.)
5. Contraindicated medications (Medical History): Gemfibrozil (inhibitor of CYP2C8) and Rifampin (inducer of CYP2C8), atorvastatin, ketoconazole, nifedipine, topiramate, and diazepam.
6. Psychiatric history:

   A) Cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires

   B) Current diagnosis of: schizophrenia or any other DSM-IV psychotic disorder, bipolar disorder, or Major Depressive Disorder (Self-Report; SCID Screen Patient Questionnaire
   * Extended (SSPQ-X))
7. Current physical dependence on alcohol or sedative-hypnotics, e.g. benzodiazepines (self-report; ASI; alcohol CAGE questions; and pattern of positive drug screens or BAL for alcohol)
8. Body Mass Index (BMI) of 40 or higher

Additional Exclusion Criteria for the fMRI portion of the Study:

Exclusion from the MRI component of the study will be based on the criteria outlined below. Participants who do not qualify or who do not agree to participate in the fMRI portion of the study will not be excluded from the main study. Exclusion criteria will be assessed during screening under NIDA-IRP screening protocol 06-DA-N415. Participants will be excluded from the fMRI portion of the study if they:

1. are left handed. Justification: Some of the neural processes assessed in this protocol may be lateralized in the brain. In order to reduce potential variance, participants will be required to be right-handed. Assessment tool(s): Edinburgh Handedness Inventory.
2. over the age of 55 years. Justification: Many cognitive processes change with age. In addition, the likelihood of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age. Therefore, older individuals, defined as those over 55, will be

   excluded from the present study.
3. have certain implanted devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts), body morphology, or claustrophobia. Justification: Implanted devices may increase the risk of MRI scanning and/or adversely affect the quality of the data; body morphology may prevent optimal positioning in the scanner and thus affect the quality of the data; participants with claustrophobia may find the MRI scan too unpleasant and may exhibit excess movement that will adversely affect the quality of the data. Assessment tool(s): Prospective participants will fill out an MRI screening questionnaire and undergo an interview with an MR technologist. Questions concerning suitability for scanning will be referred to the MR Medical Advisory Investigator. Prospective participants will be questioned about symptoms of claustrophobia and placed in the mock scanner during their first visit to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner.
4. have conditions restricting their ability to lie flat for several hours (such as coagulopathies, superficial or deep vein thrombosis, or musculoskeletal abnormalities). Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) or dangerous (e.g. familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tool(s): History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to assess comfort.
5. are cognitively impaired or learning disabled. Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited during laboratory task performance. Assessment tool(s): History of placement in special education classes as a consequence of serious learning problems and not solely as a consequence of behavioral problems, assessed during the History and Physical screening assessment.
6. have HIV or Syphilis. Justification: HIV and syphilis can each have CNS sequelae, introducing unnecessary variability into the data. Assessment tool(s): Oral HIV followed by blood test if oral test is + and Syphilis Treponemal Test (STT) without history of adequate treatment.
7. regularly use any medications that would alter CNS function, cardiovascular function, or neuronal-vascular coupling. This includes prescription medications (e.g., antidepressants, benzodiazepines, antipsychotics, anticonvulsants, barbiturates), over-the-counter medications (e.g., cold medicine), or herbal medications (e.g., Kava, Gingko biloba, St. John s wort). The only exceptions are the study medications. Justification: The use of these substances may alter the fMRI signal and/or neural functions of interest. Assessment tool(s): History and comprehensive urine drug screening to detect antidepressants, benzodiazepines, antipsychotics, anticonvulsants, and barbiturates.
8. have any current or prior neurological illnesses including, but not limited to, those listed in the main exclusion criteria. Justification: Neurological diseases alter CNS function and, possibly, the neuronal-vascular coupling that forms the basis of the fMRI signal. Assessment tool(s): History and physical examination by a qualified IRP clinician, adult ADHD Self-Report Scale, urine drug screening for anticonvulsants not disclosed by history.
9. have any other major medical condition that in the view of the investigators would compromise the integrity of the data. Justification: Many illness not explicitly covered here may alter important outcome measures. Assessment tool(s): History and physical examination by a qualified IRP clinician and CBC, urinalysis, NIDA chemistry panel (liver function tests, electrolytes, kidney function). Determination of exclusionary status will be based on laboratory values outlined in Table I for the main study, but the MAI will retain discretion to exclude participants from the fMRI/MRS secondary study based on less extreme lab results. After the screening process has been completed, the MAI will take into account all data collected in order to decide if there is an existing medical illness that would compromise participation in this research.

Additional Exclusion Criteria for the lumbar-puncture portion of the study

1. Bleeding diathesis/coagulopathy
2. Platelet count <50,000 and INR (International Normalized Ratio) greater than or equal to 1.5, or on Warfarin (coumadin)
3. Evidence of intracerebral mass based on history, neurologic exam, or papilledema on fundoscopic exam
4. Clinically significant lumbar spine disease by history, e.g. degenerative disk disease, ankylosing spondylitis or previous lumbar surgery
5. History of abnormal cranial CT scan or MRI scan, suggesting the possibility of increased intracranial pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01-04; Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

PRIMARY OUTCOMES:
Treatment response, defined as opioid abstinence without severe withdrawal symptoms during the last week of the taper (week 6) and duration in treatment (retention)

SECONDARY OUTCOMES:
Overall proportions of opioid-negative urines, proportions of participants needing adjunct medications status at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie Preston, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

REFERENCES:
- [Background] Alvarez RP, Chen G, Bodurka J, Kaplan R, Grillon C. Phasic and sustained fear in humans elicits distinct patterns of brain activity. Neuroimage. 2011 Mar 1;55(1):389-400. doi: 10.1016/j.neuroimage.2010.11.057. Epub 2010 Nov 25. PMID 21111828
- [Background] Back SE, Hartwell K, DeSantis SM, Saladin M, McRae-Clark AL, Price KL, Moran-Santa Maria MM, Baker NL, Spratt E, Kreek MJ, Brady KT. Reactivity to laboratory stress provocation predicts relapse to cocaine. Drug Alcohol Depend. 2010 Jan 1;106(1):21-7. doi: 10.1016/j.drugalcdep.2009.07.016. Epub 2009 Sep 2. PMID 19726138
- [Background] Cardenas VA, Studholme C, Gazdzinski S, Durazzo TC, Meyerhoff DJ. Deformation-based morphometry of brain changes in alcohol dependence and abstinence. Neuroimage. 2007 Feb 1;34(3):879-87. doi: 10.1016/j.neuroimage.2006.10.015. Epub 2006 Nov 28. PMID 17127079
- [Derived] Schroeder JR, Phillips KA, Epstein DH, Jobes ML, Furnari MA, Kennedy AP, Heilig M, Preston KL. Assessment of pioglitazone and proinflammatory cytokines during buprenorphine taper in patients with opioid use disorder. Psychopharmacology (Berl). 2018 Oct;235(10):2957-2966. doi: 10.1007/s00213-018-4986-5. Epub 2018 Aug 6. PMID 30079432